CLINICAL TRIAL: NCT01847209
Title: Percutaneous Image Guided Video Assisted Thoracic Surgery (VATS) Resection of Lung Lesions
Brief Title: Percutaneous Image Guided Video-Assisted Thoracic Surgery (VATS) Resection of Lung Lesions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Siemens Medical Solutions USA - CSG (Industry)
Responsible Party: Principal Investigator, Raphael Bueno, Associate Chief of Thoracic Surgery; Professor of Surgery, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012P001915
Record Dates: First submitted 2013-05-02; First posted 2013-05-06 (Estimated); Results first posted 2019-04-29 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer
Keywords: lung nodule; lung cancer; lung mass
MeSH Terms: conditions — Lung Neoplasms | interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CT Marking and VATS lung wedge resection (Experimental): Each patient with a lung nodule meeting criteria will undergo marking with fiducials followed at the same time by Video-Assisted Thoracic Surgery (VATS) lung wedge resection under CT fluoroscopy.
  Interventions: Procedure: Video-Assisted Thoracic Surgery (VATS) wedge resection

INTERVENTIONS:
Procedure: Video-Assisted Thoracic Surgery (VATS) wedge resection
  Other Names: Nodules marked with fiducials such as Kopan needles under CT fluoroscopy followed by VATS wedge resection.

SUMMARY:
This is a phase II protocol to determine the safety and feasibility of Intraoperative CT fluoroscopy guidance for lung resection for small nodules.

DETAILED DESCRIPTION:
This is a phase II protocol to determine the safety and feasibility of image guided CT marking for resection of small lung nodules. This is relevant because many such nodules are hard to localize for minimally invasive lung resection. It is hoped that this technology using fluoro CT capability available now in most operating room will improve safety and reliability of thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* peripheral lung nodules < 3cm in size
* Surgical candidate

Exclusion Criteria:

* Non surgical candidate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Bueno, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Gill RR, Zheng Y, Barlow JS, Jayender J, Girard EE, Hartigan PM, Chirieac LR, Belle-King CJ, Murray K, Sears C, Wee JO, Jaklitsch MT, Colson YL, Bueno R. Image-guided video assisted thoracoscopic surgery (iVATS) - phase I-II clinical trial. J Surg Oncol. 2015 Jul;112(1):18-25. doi: 10.1002/jso.23941. Epub 2015 May 28. PMID 26031893

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment for this study was completed in the medical clinic and started in April 2013 and included in September 2014.
Groups:
- CT Marking and VATS Lung Wedge Resection: Each patient with a lung nodule meeting criteria will undergo marking with fiducials followed at the same time by Video-Assisted Thoracic Surgery (VATS) lung wedge resection under CT fluoroscopy.
  Video-Assisted Thoracic Surgery (VATS) wedge resection
Period: Overall Study
Arm/Group | CT Marking and VATS Lung Wedge Resection
Started | 25
Completed | 23
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — No lung nodule found on intraop CT scan | 1

BASELINE CHARACTERISTICS:
Arm/Group | CT Marking and VATS Lung Wedge Resection
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 11
Age, Continuous [Median (Full Range); unit: Years] | 65 [19 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: The patient will be monitored while in the hospital by their thoracic surgical team as well as by two research nurses named Lauren Donahue, RN and Karen Magsipoc, NP. The research nurses will document any perioperative complications and mortality that arise during the patient's stay in the hospital.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | CT Marking and VATS Lung Wedge Resection
Number analyzed (Participants) | 23
Participants | 1

2. Secondary Outcome: Patients Underwent a Successful Resection
Description: Number of patients who underwent a successful resection which is measured by an accurate and appropriate resection in a given timeline
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | CT Marking and VATS Lung Wedge Resection
Number analyzed (Participants) | 23
Participants | 23

ADVERSE EVENTS:
Time Frame: 1 year from consent and surgery
Arm/Group | CT Marking and VATS Lung Wedge Resection
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 1/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CT Marking and VATS Lung Wedge Resection (N=23)
Received increased radiation dose (Surgical and medical procedures) | 1 (1) — Patient received an increase dose of radiation than what was estimated in the protocol. The dose given to the patient is not dangerous and is equivalent to 2-3 CT scans The patient has done well and has had no adverse effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-01-29): https://cdn.clinicaltrials.gov/large-docs/09/NCT01847209/Prot_SAP_000.pdf
  • Informed Consent Form (2013-07-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT01847209/ICF_001.pdf